CLINICAL TRIAL: NCT05211271
Title: Evaluating Thermal Ablation in the Treatment of Cervical Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Kamenge University Hospital, Burundi University, Burundi (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM/CE/05/08/2018
Record Dates: First submitted 2021-12-02; First posted 2022-01-27 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2022-01

CONDITIONS: Cervical Neoplasia
Keywords: cervical neoplasia; treatment; thermal ablation; longitudinal study; LMIC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Treatment of cervical neoplasia by thermal ablation
  Interventions: Device: Treatment of cervical neoplasia by thermal ablation

INTERVENTIONS:
Device: Treatment of cervical neoplasia by thermal ablation — Women screened for cervical cancer by visual inspection with diluted acetic acid (VIA) presenting lesions eligible for ablative treatment were treated by thermal ablation. The treatment consisted in applying the probe on the lesion for 45 seconds at 100 degrees Celsius, with one to up to five applications depending on the lesion size. Following treatment, women were inquired about the pain level during the procedure, their satisfaction level of the procedure and whether they would recommend this treatment to their relatives. Women had a follow-up visit at 6 weeks to assess any complication of the procedure. Women were rescreened at 12 months, to evaluate the cure rate and any long-term adverse events.

SUMMARY:
Longitudinal study in Burundi to evaluate the effectiveness, the acceptability and safety of thermal ablation in the treatment of cervical neoplasia.

DETAILED DESCRIPTION:
The study population consisted of women with an abnormal VIA test or an abnormal colposcopy examination. A total of 86 women with lesions eligible to ablative treatment were counselled and treated by thermal ablation. Informed consent was signed by each participant. Just after treatment, they were inquired about the level of pain during the procedure, and their level of satisfaction with the treatment. They were followed-up at 6 weeks for any complication and re-assessed by VIA and colposcopy at 12 months for any persistent or recurrent lesion and for any adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Women residing in Burundi and referred to the tertiary hospital after a positive VIA test

Exclusion Criteria:

* Lesion occupying the 4 quadrants of the cervix
* Not visible squamous columnar junction (not Type 1 TZ)
* Vaginal or endocervical lesion
* Lesion subjective of cervical cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Cure rate based on VIA and colposcopy assessment | 1 year
  Effectiveness is measured by the cure rate after 1 year based on VIA and colposcopy assessment.
Acceptability of thermal ablation | 6 weeks
  Measured by existence of minor/moderate adverse events during the follow-up.
Acceptability of thermal ablation | At day 1
  Measured by the satisfaction level using a nine-level Likert scale (from 1. Very unsatisfied to 9. very satisfied).
Safety of thermal ablation | 1 year
  Measured by existence of severe adverse events during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvestre Bazikamwe, MD, Principal Investigator — Kamenge University Hospital, Burundi University, Bujumbura, Burundi; Catherine Sauvaget, MD, PhD, Principal Investigator — International Agency for Research on Cancer
Locations (1):
- Kamenge University Hospital, Bujumbura, Burundi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sauvaget C, Bazikamwe S, Lucas E, Ndayikengurukiye A, Harerimana S, Barango P. Evaluation of effectiveness, acceptability and safety of thermal ablation in the treatment of cervical neoplasia in Burundi. Int J Cancer. 2022 Oct 1;151(7):1120-1126. doi: 10.1002/ijc.34117. Epub 2022 Jun 3. PMID 35567576